CLINICAL TRIAL: NCT03275922
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Study To Evaluate The Efficacy And Safety Of Zolmitriptan Nasal Spray For The Treatment Of Acute Migraine In Subjects Ages 6 To 11 Years, With An Open-Label Extension
Brief Title: Efficacy & Safety Of Zomig Nasal Spray For Acute Migraine Treatment In Subjects 6 To 11 Years, With OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX229-B16-01
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-07

CONDITIONS: Migraine
Keywords: Migraine; Headache; Pain; Efficacy; Pediatric
MeSH Terms: conditions — Migraine Disorders; Headache; Pain

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Double-blind, Placebo-controlled, Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Run-in - ZNS - Placebo - OLE (Other): After Run-in period, subjects will be randomized to ZNS followed by placebo ZNS. Upon successful completion of Part 1, subjects may enroll into OLE (Part 2).
  Interventions: Drug: Placebo ZNS; Drug: ZNS
- Run-in - Placebo - ZNS - OLE (Other): After Run-in period, subjects will be randomized to placebo ZNS followed by ZNS. Upon successful completion of Part 1, subjects may enroll into OLE (Part 2).
  Interventions: Drug: Placebo ZNS; Drug: ZNS

INTERVENTIONS:
Drug: Placebo ZNS — Placebo Zolmitriptan Nasal Spray
  Other Names: Placebo
Drug: ZNS — Zolmitriptan Nasal Spray

SUMMARY:
To evaluate the efficacy and safety of zolmitriptan nasal spray (ZNS) in the acute treatment of migraine headache in subjects ages 6 to 11 years.

Part 1: Approximately 20 weeks (includes screening and double-blind treatment).

* Screening will be performed based on the inclusion exclusion criteria specified in the study protocol.
* Randomize approximately 288 subjects into the double-blind crossover phase.

Part 2: Approximately 100 subjects who complete the double-blind crossover phase will enter part 2, a 6 month open-label safety extension (OLE).

Efficacy will be evaluated in the double-blind part of the trial. Safety will be evaluated in both the double-blind and the OLE.

ELIGIBILITY:
Inclusion Criteria

1. Parent or legal guardian is able to provide written informed consent and subject is able to provide assent.
2. Subjects ages 6 to 11 years throughout the double-blind portion of the studyAn established diagnosis of migraine
3. By history, average migraine frequency of ≥ 2 attacks per month lasting on average ≥ 3 hours per attack
4. By history, experiences at least 16 headache-free days per month on average

Exclusion Criteria:

1. History of ischemic or vasospastic heart disease, arrhythmias associated with accessory conduction pathways (eg, Wolff-Parkinson-White syndrome), cerebrovascular disease, hemiplegic or basilar artery migraine, peripheral vascular disease, ischemic bowel disease, uncontrolled hypertension, recent (within 24 hours) or use of another 5HT1 agonist, ergots or ergotamine-containing medications.
2. Any medical condition, including severe hepatic impairment, which, in the opinion of the investigator, may put the subject at increased risk with exposure to zolmitriptan, or may interfere with the safety or efficacy assessments.
3. Had an unacceptable adverse experience following previous use of any 5HT1B/1D agonist drug (in the opinion of the investigator).
4. Had not experienced satisfactory relief from migraine pain during prior treatment with 2 or more adequate courses of triptans.
5. Prior use of any nasal spray (triptan or dihydroergotamine [DHE]) for the acute treatment of migraine
6. Disease or anatomic abnormalities of the nasal cavity precluding or complicating the use of ZNS.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 374 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Pain-free status at 2 hours post treatment | 2 hours post-dose
  Headache pain intensity is assessed by the subjects immediately prior to treatment and 2 hours post-dose using a 4-point headache pain intensity scale (severe = 3, moderate = 2, mild = 1, or none = 0).

SECONDARY OUTCOMES:
Proportion of subjects who achieve pain-free status at 24 hours post-dose | 24 hours post-dose
  The headache pain intensity is assessed by the subjects using a 4-point headache pain intensity scale (severe = 3, moderate = 2, mild = 1, or none = 0).
Headache response at 24 hours post-dose | 24 hours post-dose
  The subject diary captures the headache severity using a 4-point headache pain intensity scale (severe = 3, moderate = 2, mild = 1, or none = 0). Headache response is defined as a reduction in moderate (2) or severe (3) pain to mild (1) or no (0) pain at 24 hour post-dose.
Sustained headache response at 24 hours post-dose | 24 hours post-dose
  Sustained headache response is defined as a reduction in migraine headache pain intensity from severe or moderate to mild or none at 2 hours which is then maintained (without a return to moderate or severe pain) at 24 hours with no use of rescue medication prior to the 24 hour assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (47):
- United States (47):
  - Phoenix Children's Hospital (149), Phoenix, Arizona
  - Arkansas Children's Hospital (109), Little Rock, Arkansas
  - Advanced Research Center, Inc (134), Anaheim, California
  - Sierra Medical Research (124), Fresno, California
  - Shailesh M. Asaikar, MD. Inc. DBA Child and Adolescent Neurology Consultatns (119), Sacramento, California
  - Children's Hospital Colorado (154), Aurora, Colorado
  - Blue Sky Neurology (106), Englewood, Colorado
  - IMMUNOe Research Centers (150), Thornton, Colorado
  - Ki Health Partners, LLC dba New England INstitute for Clinical Research (128), Stamford, Connecticut
  - Children's National Health System (141), Washington D.C., District of Columbia
  - NW Florida Clinical Research Group, LLC (122), Gulf Breeze, Florida
  - Clinical Neuroscience Solutions, Inc. (127), Jacksonville, Florida
  - Axcess Medical Research (126), Loxahatchee Groves, Florida
  - Biotech Pharmaceutical Group (138), Miami, Florida
  - Sanitas Medical and Dental Institute/dba Sanitas Research, LLC (142), Miami, Florida
  - Laszlo J. Mate, M.D., P.A. (153), North Palm Beach, Florida
  - Clincial Neuroscience Solutions, Inc. (136), Orlando, Florida
  - Pediatric Neurology, PA (125), Orlando, Florida
  - East Florida Research (143), Port Saint Lucie, Florida
  - Pedatric Epilepsy & Neurology Specialists (157), Tampa, Florida
  - Premiere Research Institute @ Palm Beach Neurology, PA (105), West Palm Beach, Florida
  - Clinical Integrative Research Center of Atlanta (121), Atlanta, Georgia
  - NuDirections Clinical Research, LLC (159), Atlanta, Georgia
  - iResearch Atlanta, LLC (146), Decatur, Georgia
  - Meridian Clinical Research, LLC (130), Savannah, Georgia
  - Josephson Wallack Munshower Neurology P.C. (114), Indianapolis, Indiana
  - Kosair Charities Pediatric Clinical Research Unit (120), Louisville, Kentucky
  - Michigan Head-Pain and Neurological Institute (103), Ann Arbor, Michigan
  - Mercy Research (116), St Louis, Missouri
  - Clinical Research Center of NJ (123), Voorhees Township, New Jersey
  - Dent Neurosciences Research Center (129), Amherst, New York
  - OnSite Clinical Solutions, LLC (155), Charlotte, North Carolina
  - Headache Wellness Center (Site 152), Greensboro, North Carolina
  - Raleigh Neurology Associates, PA (113), Raleigh, North Carolina
  - Akron Children's Hospital (site 139), Akron, Ohio
  - Cincinnati Children's Hospital (140), Cincinnati, Ohio
  - Preferred Primary Care Physicians, Inc. (115), Pittsburgh, Pennsylvania
  - Access Clinical Trials, Inc. (151), Nashville, Tennessee
  - Texas Neurology, P.A. (110), Dallas, Texas
  - Children's Medical Center Dallas (147), Dallas, Texas
  - J. Lewis Research Inc. Foothill Family Clinic (107), Salt Lake City, Utah
  - Primary Children's Hospital Outpatient Services (117), Salt Lake City, Utah
  - Granger Medical Holladay (111), Salt Lake City, Utah
  - Pediatric Research of Charlottesville, LLC (104), Charlottesville, Virginia
  - Northwest Clinical Research Center (132), Bellevue, Washington
  - Multicare Health System- Mary Bridge Pediatrics- Tacoma (158), Tacoma, Washington
  - Marshfield Clinic (145), Marshfield, Wisconsin